CLINICAL TRIAL: NCT05735964
Title: Indocyanine Green (ICG) and Near Infrared Fluorescence (NIRF) Guided Assessment of the Bowel and Oesophageal Anastomosis During Repair of Oesophageal Atresia with Distal Trachea-oesophageal Fistula (OA/dTOF): a Cohort Pilot Study
Brief Title: Use of Indocyanine Green During Primary Repair of Oesophageal Atresia and Distal Tracheo-oesophageal Fistula
Acronym: iTOF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Birmingham Women's and Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22/BC/ONC/NO/633
Record Dates: First submitted 2022-12-20; First posted 2023-02-21 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-08

CONDITIONS: Tracheo-Esophageal Fistula with Atresia of Esophagus
MeSH Terms: conditions — Esophageal atresia with or without tracheoesophageal fistula | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: Consecutive patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ICG (Experimental): Patients in this single arm will receive ICG during their surgery
  Interventions: Drug: Indocyanine green

INTERVENTIONS:
Drug: Indocyanine green — Intravenous and endoluminal dosing

SUMMARY:
This study aims to look at babies having a primary or delayed primary oesophageal repair for OA with dTOF to evaluate if using Indocyanine green (ICG) and near infrared fluorescence (NIRF) can decrease the rates of anastomotic leaks and/or predict which patients they will happen in. The latter evaluation would help counsel parents and mean that further research can evaluate if other tactics can prevent the leak being a moderate or severe problem. These may include, but not be limited to, extra anastomotic sutures, insertion of a chest drain at the time of surgery (if this had not previously been considered) delaying oral feeding or using medications to dry up the saliva prophylactically (these medications have been shown to reduce the length of time it takes leaks to seal). Any technique that can reduce leak rates in oesophageal atresia is to be welcomed.

Additionally ICG may artifactually affect both peripheral oxygen readings (cause a transient decrease) and cerebral near infrared spectroscopy (NIRS) values (cause a transient increase). This is due to the temporary, dose dependent, interference of the dye with the mechanism of action of the monitoring rather than a physiological effect on oxygen levels. To date there has been no study investigating the effects of ICG on oxygen saturation and cerebral NIRS in neonates undergoing OA and/or dTOF repair.

The theory is an extension from adult practice following oesophagectomy for cancer where there was a reduction in anastomotic leaks when using ICG/NIRF perfusion assessment. Another study in bariatric surgery using an enteral ICG/NIRF assessment was highly sensitive for anastomotic leaks allowing management of them intra-operatively.

Objectives are to

1. Identify if the appearances of ICG/NIRF can predict anastomotic leaks
2. Identify if the ICG/NIRF images would engender a change in operative management leading to a reduced leak rate
3. Give a detailed report on the effects of ICG on oxygen readings This would be a cohort pilot study of 20 patients with the aim of informing a subsequent multi-centre Randomised controlled trial

DETAILED DESCRIPTION:
Anastomotic leaks can have wide ranging consequences. If they can be predicted and/or prevented clinical outcomes for patients would be improved along with shorter length of stay and reduced cost to the national health service (NHS) in the short, medium, and long term. These patients would require less bed days both on inpatient wards and paediatric intensive care units enabling the management of other children.

This study will evaluate if ICG/NIRF tissue perfusion diagnostics can show if the fistula (distal oesophagus) end is ischaemic (has poor blood flow) prior to anastomosis. Ischaemic ends are well recognised to relate to leakage although in OA the role of mucosal apposition is poorly understood. This intervention would afford the operator the opportunity to perform a fully vascularised join if feasible and also indicate if ischaemia predicts anastomotic leaks.

It will also evaluate if post-anastomosis intravenous and enteral dosing of ICG with NIRF assessment is able to predict those who will suffer from a leak whether that be clinical or radiological.

There is little data on the effect of ICG on peripheral oxygen saturation readings, or of its effect on near infrared spectroscopy readings in neonates. This study will record the effects on peripheral saturation and near-infrared spectroscopy readings which are used routinely in babies having this type of surgery. It will compare these readings to arterial blood oxygenation readings from a blood gas analyser. Blood gases are routinely taken during this procedure and so this will not involve any extra blood testing over and above what is ordinarily performed.

ELIGIBILITY:
Inclusion Criteria:

Pre-operative

* Diagnosis of oesophageal atresia with distal trachea-oesophageal fistula (OA/dTOF)
* Plan for primary or delayed primary oesophageal anastomosis

Intra-operative

* Diagnosis of OA/dTOF confirmed by standard methods
* Primary or delayed primary oesophageal anastomosis considered clinically, physiologically, and technically feasible

Exclusion Criteria:

Pre-operative

* Under 2.5kg in weight
* Complex cardiac disease
* Allergic to ICG
* Allergic to iodine or iodides
* Hyperthyroidism
* Chronic Kidney Disease stage V
* Unwilling to participate
* Those in whom exchange transfusion is indicated due to hyperbilirubinemia

Intra-operative

• Anaesthetic concerns contra-indicating the use of intravenous ICG due its temporary effect on oxygen saturation readings prior to injection of ICG

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Intravenous ICG | Within two weeks of surgery
  Number of patients with abnormal perfusion will have a clinical and/or radiological anastomotic leak
Enteral ICG | Within two weeks of surgery
  Number of patients in whom ICG given enterally shows an anastomotic leak

SECONDARY OUTCOMES:
Delphi | Within a year following surgery
  Number of patients in whom ICG given prior to anastomosis causes a change in intra-operative plan
Peripheral oxygen saturations (SpO2) | Within a year following surgery
  In how many patients does the intravenous injection of ICG alter the peripheral oxygenation and/or near infrared spectroscopy readings.

CONTACTS AND LOCATIONS:
Overall Officials: Max Pachl, Principal Investigator — Birmingham Women's and Children's NHS Foundation Trust, UK
Locations (1):
- Birmingham children's hospital, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
data used in publications will be shared in peer-reviewed literature

REFERENCES:
- [Background] Kalmar CL, Reed CM, Peery CL, Salzberg AD. Intraluminal indocyanine green for intraoperative staple line leak testing in bariatric surgery. Surg Endosc. 2020 Sep;34(9):4194-4199. doi: 10.1007/s00464-020-07606-4. Epub 2020 May 8. PMID 32385707
- [Background] Schmedding A, Wittekindt B, Schloesser R, Hutter M, Rolle U. Outcome of esophageal atresia in Germany. Dis Esophagus. 2021 Apr 7;34(4):doaa093. doi: 10.1093/dote/doaa093. PMID 32995846
- [Background] Long AM, Tyraskis A, Allin B, Burge DM, Knight M. Oesophageal atresia with no distal tracheoesophageal fistula: Management and outcomes from a population-based cohort. J Pediatr Surg. 2017 Feb;52(2):226-230. doi: 10.1016/j.jpedsurg.2016.11.008. Epub 2016 Nov 13. PMID 27894760
- [Background] Burge DM, Shah K, Spark P, Shenker N, Pierce M, Kurinczuk JJ, Draper ES, Johnson PR, Knight M; British Association of Paediatric Surgeons Congenital Anomalies Surveillance System (BAPS-CASS). Contemporary management and outcomes for infants born with oesophageal atresia. Br J Surg. 2013 Mar;100(4):515-21. doi: 10.1002/bjs.9019. Epub 2013 Jan 18. PMID 23334932
- [Background] Allin B, Knight M, Johnson P, Burge D; BAPS-CASS. Outcomes at one-year post anastomosis from a national cohort of infants with oesophageal atresia. PLoS One. 2014 Aug 25;9(8):e106149. doi: 10.1371/journal.pone.0106149. eCollection 2014. PMID 25153838
- [Background] Comella A, Tan Tanny SP, Hutson JM, Omari TI, Teague WJ, Nataraja RM, King SK. Esophageal morbidity in patients following repair of esophageal atresia: A systematic review. J Pediatr Surg. 2021 Sep;56(9):1555-1563. doi: 10.1016/j.jpedsurg.2020.09.010. Epub 2020 Sep 19. PMID 33051081
- [Background] Weber F, Scoones GP. A practical approach to cerebral near-infrared spectroscopy (NIRS) directed hemodynamic management in noncardiac pediatric anesthesia. Paediatr Anaesth. 2019 Oct;29(10):993-1001. doi: 10.1111/pan.13726. Epub 2019 Aug 29. PMID 31437328
- [Background] Bishay M, Giacomello L, Retrosi G, Thyoka M, Nah SA, McHoney M, De Coppi P, Brierley J, Scuplak S, Kiely EM, Curry JI, Drake DP, Cross KM, Eaton S, Pierro A. Decreased cerebral oxygen saturation during thoracoscopic repair of congenital diaphragmatic hernia and esophageal atresia in infants. J Pediatr Surg. 2011 Jan;46(1):47-51. doi: 10.1016/j.jpedsurg.2010.09.062. PMID 21238638
- [Background] Stolwijk LJ, van der Zee DC, Tytgat S, van der Werff D, Benders MJNL, van Herwaarden MYA, Lemmers PMA. Brain Oxygenation During Thoracoscopic Repair of Long Gap Esophageal Atresia. World J Surg. 2017 May;41(5):1384-1392. doi: 10.1007/s00268-016-3853-y. PMID 28058473
- [Background] Baek HY, Lee HJ, Kim JM, Cho SY, Jeong S, Yoo KY. Effects of intravenously administered indocyanine green on near-infrared cerebral oximetry and pulse oximetry readings. Korean J Anesthesiol. 2015 Apr;68(2):122-7. doi: 10.4097/kjae.2015.68.2.122. Epub 2015 Mar 30. PMID 25844129
- [Background] De Gasperi A, Mazza E, Prosperi M. Indocyanine green kinetics to assess liver function: Ready for a clinical dynamic assessment in major liver surgery? World J Hepatol. 2016 Mar 8;8(7):355-67. doi: 10.4254/wjh.v8.i7.355. PMID 26981173
- [Background] Kulshrestha S, Kulshrestha M, Tewari V, Chaturvedi N, Goyal A, Sharma RK, Sarkar D, Tandon JN, Katyal V. Conservative Management of Major Anastomotic Leaks Occurring after Primary Repair in Esophageal Atresia with Fistula: Role of Extrapleural Approach. J Indian Assoc Pediatr Surg. 2020 May-Jun;25(3):155-162. doi: 10.4103/jiaps.JIAPS_73_19. Epub 2020 Apr 11. PMID 32581443
- [Background] Cui X, He Y, Chen L, Lin Y, Zhang J, Zhou C. The Value of Thoracic Lavage in the Treatment of Anastomotic Leakage After Surgery for Type III Esophageal Atresia. Med Sci Monit. 2020 Mar 11;26:e919962. doi: 10.12659/MSM.919962. PMID 32158013
- [Background] Campos J, Tan Tanny SP, Kuyruk S, Sekaran P, Hawley A, Brooks JA, Bekhit E, Hutson JM, Crameri J, McLeod E, Teague WJ, King SK. The burden of esophageal dilatations following repair of esophageal atresia. J Pediatr Surg. 2020 Nov;55(11):2329-2334. doi: 10.1016/j.jpedsurg.2020.02.018. Epub 2020 Feb 19. PMID 32143903
- [Background] Donoso F, Hedenstrom H, Malinovschi A, E Lilja H. Pulmonary function in children and adolescents after esophageal atresia repair. Pediatr Pulmonol. 2020 Jan;55(1):206-213. doi: 10.1002/ppul.24517. Epub 2019 Sep 18. PMID 31535483
- [Background] Guillen G, Lopez-Fernandez S, Molino JA, Bueno J, Lopez M. [Pilot experience with indocyanine green navigation in pediatric surgery]. Cir Pediatr. 2019 Jul 29;32(3):121-127. Spanish. PMID 31486303
- [Background] Oetzmann von Sochaczewski C, Heimann A, Linder A, Kempski O, Muensterer OJ. Esophageal Blood Flow May Not Be Directly Influenced by Anastomotic Tension: An Exploratory Laser Doppler Study in Swine. Eur J Pediatr Surg. 2019 Dec;29(6):516-520. doi: 10.1055/s-0038-1676979. Epub 2019 Jan 4. PMID 30609438
- [Background] Petit LM, Righini-Grunder F, Ezri J, Jantchou P, Aspirot A, Soglio DD, Faure C. Prevalence and Predictive Factors of Histopathological Complications in Children with Esophageal Atresia. Eur J Pediatr Surg. 2019 Dec;29(6):510-515. doi: 10.1055/s-0038-1676505. Epub 2018 Dec 19. PMID 30566986
- [Background] Vergouwe FW, Gottrand M, Wijnhoven BP, IJsselstijn H, Piessen G, Bruno MJ, Wijnen RM, Spaander MC. Four cancer cases after esophageal atresia repair: Time to start screening the upper gastrointestinal tract. World J Gastroenterol. 2018 Mar 7;24(9):1056-1062. doi: 10.3748/wjg.v24.i9.1056. PMID 29531469
- [Background] Agzarian J, Visscher SL, Knight AW, Allen MS, Cassivi SD, Nichols FC 3rd, Shen KR, Wigle D, Blackmon SH. The cost burden of clinically significant esophageal anastomotic leaks-a steep price to pay. J Thorac Cardiovasc Surg. 2019 May;157(5):2086-2092. doi: 10.1016/j.jtcvs.2018.10.137. Epub 2018 Nov 15. PMID 30558876